CLINICAL TRIAL: NCT03714100
Title: Use of Tele-Exercise as an Alternative Delivery Channel for Translating an Evidence-Based Fall-Prevention Program Into Practice for Older Adults in West Virginia
Brief Title: Use of Tele-Exercise for Translating an Evidence-Based Fall-Prevention Program for Older Adults in West Virginia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Dina L Jones, PT, PhD, Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3R49CE002109-05S1 (NIH)
Record Dates: First submitted 2018-10-11; First posted 2018-10-22 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Accidental Falls
MeSH Terms: interventions — Tai Ji; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MFBB intervention (Experimental): All participants will attend Tai Ji Quan: Moving for Better Balance classes twice a week for 16 weeks. Groups of participants will gather at a local community site that has videoconferencing capabilities. The instructor will be teaching the class from a different location via a live video feed.
  Interventions: Behavioral: Tai Ji Quan: Moving for Better Balance

INTERVENTIONS:
Behavioral: Tai Ji Quan: Moving for Better Balance — Participants will attend one-hour Tai Ji Quan: Moving for Better Balance classes twice a week for 16-weeks. Groups of participants will gather at a local community site that has videoconferencing capabilities. The instructor will be teaching the class from a different location via a live video feed.
  Other Names: Tai Chi, Physical Activity, Exercise

SUMMARY:
West Virginia (WV) has a critical need for resources to reach more of its older adults with fall-prevention programming. The Tai Ji Quan: Moving for Better Balance® (TJQMBB) program is an evidence-based, Centers for Disease Control and Prevention (CDC)-approved, community-delivered, physical activity fall-prevention intervention for older adults. The program is efficacious and effective in reducing falls in older adults, and has been translated into clinical and community settings. Programs delivered in one setting; however, may not automatically translate to others.

Using telehealth technology to deliver exercise classes (i.e. tele-exercise) is one alternative to the traditional, face-to-face, group exercise classes where the instructor and participants are in the same room. We propose delivering tele-TJQMBB to older adults using a computer, television, and the internet. This delivery mode will allow us to recruit instructors from any location (e.g., urban areas), and with possibly more experience, yet still reach older adults in communities without instructors.

DETAILED DESCRIPTION:
West Virginia (WV) has a critical need for resources to reach more of its older adults with fall-prevention programming. The Tai Ji Quan: Moving for Better Balance® (TJQMBB) program is an evidence-based, CDC-approved, community-delivered, physical activity fall-prevention intervention for older adults. The program is efficacious and effective in reducing falls in older adults, and has been translated into clinical and community settings. Programs delivered in one setting; however, may not automatically translate to others. We recently completed a CDC-funded study which successfully translated a 16-week TJQMBB intervention into 20 faith-based organizations in 7 rural WV counties. In the maintenance phase of the study (i.e., post intervention), only 38% of classes continued despite the fact that 87% of participants expressed a desire to continue. The rate limiting factor for continuing classes in these rural areas was lack of instructors. Thus, there is a vital need to further translate TJQMBB into practice using alternative delivery channels to increase the reach and maintenance of the program, especially in rural areas where instructors are less available.

Using telehealth technology to deliver exercise classes (i.e. tele-exercise) is one alternative to the traditional, face-to-face, group exercise classes where the instructor and participants are in the same room. We propose delivering tele-TJQMBB to older adults using a computer, television, and the internet. This delivery mode will allow us to recruit instructors from any location (e.g., urban areas), and with possibly more experience, yet still reach older adults in communities without instructors.

The purpose of this translational study is to work with our injury control, technology, and wellness partners to: 1) implement a 16-week intervention of the tele-TJQMBB classes in 120 older adults at 12 community sites in 4 WV counties; 2) describe functional, self-reported, and fall/injury outcomes; and 3) evaluate the translation of tele-TJQMBB with respect to its Reach into the target population (number of participants), Effectiveness (participant outcomes), Adoption (number of sites, instructors, classes), Implementation (fidelity ratings), and Maintenance (satisfaction, continued participation) using the Re-aim Framework. Demonstrating that tele-TJQMBB is effective would provide an additional delivery channel for the program, help overcome the barrier of identifying instructors in rural areas, and in the future, allow for the number of classes to be expanded to reach more older adults, provide more community-based programs in which to refer older adults to, and enhance overall maintenance of the program. To our knowledge, this is the first study to translate an evidence-based, group, fall-prevention exercise program using an alternative delivery method in a priority population, and thus, may serve as a model for reaching other underserved older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 55 and older
* Community-dwelling
* Able to attend 2, 1-hour Tai Ji Quan: Moving for Better Balance classes a week for 16 weeks
* Able to attend 2 testing sessions for data collection (Testing sessions will be scheduled the week before classes begin and the week after the classes end)
* Able to walk at least 2 city blocks with or without an assistive device

Exclusion Criteria:

* Lack reliable transportation
* Unable to speak English

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Four Square Test | At 16 weeks after start of intervention
  Balance will be assessed using the Four Square Test which requires participants to step over low objects and move in 4 directions.

SECONDARY OUTCOMES:
Gait Speed: 5-meter walk test | Collected at end of the intervention (16 weeks)
  A self-selected walking speed will be used to measure gait speed.
Mobility: Timed up-and-go test | Collected at end of the intervention (16 weeks)
  A participant stands from a chair, walks 3 meters at a self-selected pace, turns, and returns to the chair to sit.
Lower extremity strength: 5-chair stands test | Collected at end of the intervention (16 weeks)
  A participant is times as they stand up from a seated position five times. The test ends when the participant achieves the standing position on the 5th repetition.
Physical Activity: National Health Interview Survey (NHIS) | Collected at end of the intervention (16 weeks)
  2016 NHIS questions
Health-related quality of life: Short Form-12 (SF-12) | Collected at end of the intervention (16 weeks)
  Questionnaire used to measure functional health and well-being from the participant's point of view.
Fear of falling: Falls Efficacy Scale | Collected at end of the intervention (16 weeks)
  Tool that measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity.
Fall frequency (falls, fallers, and frequent fallers) | Collected at end of the intervention (16 weeks)
  Participants will be given a monthly calendar with a pre-paid postage return envelope to record falls/injuries.
Fall rates (falls/person-months) | Collected at baseline, at the end of the intervention (16 weeks), and 32 weeks after the start of the study
  Participants will be given a monthly calendar with a pre-paid postage return envelope to record falls/injuries.
Injury frequency | Collected at end of the intervention (16 weeks)
  Participants will be given a monthly calendar with a pre-paid postage return envelope to record falls/injuries.
Injury severity | Collected at end of the intervention (16 weeks)
  If an injury was reported on the falls calendar, we will conduct a telephone interview with the participant to obtain the mechanism of the fall, the type and severity of any injuries, and details about any medical care that was received.
Medical care received | Collected at end of the intervention (16 weeks)
  If an injury was reported on the falls calendar, we will conduct a telephone interview with the participant to obtain the mechanism of the fall, the type and severity of any injuries, and details about any medical care that was received.
Process outcomes | Collected at end of intervention (16 weeks)
  Exercise adherence and adverse events will be collected via attendance and injury forms

CONTACTS AND LOCATIONS:
Overall Officials: Dina L Jones, PT, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No